CLINICAL TRIAL: NCT03558022
Title: Vascular Responses to Sympathetic Activation and Altered Shear Rate: The Impact of Hypertension and Sodium Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20013060
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salt Pills (Experimental): One week on low salt diet plus salt pills
  Interventions: Dietary Supplement: Salt Pills
- Placebo Pills (Placebo Comparator): One week on low salt diet plus placebo pills
  Interventions: Dietary Supplement: Placebo Pills

INTERVENTIONS:
Dietary Supplement: Salt Pills — 7 days of a low sodium diet plus 4 salt pills (sodium chloride) taken 3 times daily with meals (approximately 7000 milligrams per day)
  Arms: Salt Pills
Dietary Supplement: Placebo Pills — 7 days of low sodium diet plus 4 placebo pills (microcrystalline cellulose) taken 3 times daily with meals
  Arms: Placebo Pills

SUMMARY:
The aim of this study is to determine if alterations in sodium intake alter peripheral vascular function and exercise tolerance in young individuals.

DETAILED DESCRIPTION:
Sodium intake is a major contributor to the development of hypertension in the developed world. Interestingly, it has been recently revealed that, in addition to the cardiovascular dysfunction associated with high sodium intake-induced hypertension, individuals who have unaltered blood pressure after chronic high sodium intake, termed salt resistant, report similar reductions in cardiovascular function when compared to salt sensitive individuals. While the extent to which this high sodium intake negatively alters cardiovascular structure as well as function is currently being explored, little is known about how high sodium intake impacts vascular function and blood flow regulation during exercise. Therefore, this study will determine if alterations in sodium intake alter peripheral vascular function and exercise tolerance in young individuals. The investigators hypothesize that increases in sodium intake will reduce exercise-induced arterial dilation in response to shear and result in exercise intolerance, via impaired functional sympatholysis, at moderate-to-high exercise workloads. Furthermore, the investigators hypothesize that these changes in blood flow regulation and exercise tolerance in young individuals will be reversed following antioxidant supplementation, implicating the role of oxidative stress in this dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* normotensive blood pressure (Systolic <120 AND Diastolic <80
* free of cardiovascular disease and any evidence of thyroid, renal, metabolic, pulmonary or neurological disease
* non-obese (BMI <30 and/or Body fat < 25% for men, and < 30% for women)
* no tobacco use
* no medications that could affect vascular function or oxidative stress
* not sedentary

Exclusion Criteria:

* individual with cardiovascular, pulmonary, or metabolic disease or taking medications that may alter cardiovascular, pulmonary, or metabolic function
* subjects will be asked to maintain a dietary record for one week subsequent to the pre-screening and if this reveals a diet that differs substantially from the "typical" average diet, the subject will not be eligible
* subjects will be excluded from the study if dietary records reveal significant caloric restriction and/or vitamin/mineral deficiencies
* pregnant women, prisoners, and children will not be eligible for this study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Arterial Dilation in Response to Exercise | After 7 day high salt supplementation vs After 7 day low salt supplementation
  Percent change is arterial diameter when compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Garten, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States